CLINICAL TRIAL: NCT02322554
Title: The Registry of Cellular and Tissue Based Therapies for Chronic Wounds and Ulcers
Brief Title: Cellular and Tissue Based Therapy Registry
Acronym: CTPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: U.S. Wound Registry (Other)
Responsible Party: Sponsor
Other Study IDs: CDR002
Record Dates: First submitted 2014-11-23; First posted 2014-12-23 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Foot Ulcers; Venous Stasis Ulcer; Pressure Ulcer; Chronic Non Healing Wound; Surgical Wound Dehiscence
Keywords: electronic health records; Qualified Clinical Data Registry; PQRS; quality reporting; cellular based products; bioengieered skin; USWR
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer; Surgical Wound Dehiscence | interventions — Cell Count; Apligraf; TransCyte; poly(divinyl-co-N-vinylpyrrolidinone); Alloderm; integra artificial skin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- wounds treated with CTPs: All cellular and tissue based products currently reimbursed in the hospital based outpatient department, administered at intervals as determined in the course of clinical practice
  Interventions: Biological: Cellular and tissue based products

INTERVENTIONS:
Biological: Cellular and tissue based products — Procedure: Application of device or biological to wounds
  Other Names: Apligraf; Dermagraft; Epifix; Oasis; Talymed; Primatrix; Theraskin; Grafix; Dermaspan; Alloderm; Amnioband; GraftJacket; Integra; Matristem

SUMMARY:
The goal of the Cellular and Tissue Based Therapy Registry (CTPR) for Wounds is to provide real world patient data from electronic health records submitted to meet Stage 2 Meaningful Use in order to understand the value of these products among patients with chronic wounds and ulcers. Randomized, controlled trials to establish product efficacy routinely exclude patients with the co-morbid conditions common to patients seen in usual clinical practice and thus the results of these RCTs tend to be non-generalizable. Little is known about the effectiveness of CTPs among typical patients.

DETAILED DESCRIPTION:
The goal of the Cellular and Tissue Based Therapy Registry (CTPR) for Wounds is to provide comparative effectiveness data for patients with chronic wounds and ulcers and to understand whether clinical practice guidelines are followed in the use of these products. These products are referred to by a variety of names of which are inaccurate reflections of their structure or purpose (e.g. Cellular and Engineered Tissue Alternatives, "bioengineered tissues," "biological dressings"). The preferred term is cellular and/or tissue based products (CTPs). CTPs are utilized for their biological influence on the healing process by stimulating or supporting healing. They may or may not be incorporated into regenerating tissue. Both tissue derived and biosynthetic products may be made with or without dead cells and biomaterials made of living cells may be comprised of autologous cells (cultured and not cultured), xenogenic, or allogenic cells (minimally manipulated, cultured, immortal).The diversity of products and the rate at which they are becoming available for clinical use make it impossible to perform randomized controlled trials to compare their effectiveness against one another. Effectiveness in real world patients is the best current option to understand the role of CTPs in wound healing.

Hospital based outpatient wound centers participating in the US Wound Registry agree to provide data as part of quality initiatives and to meet their Stage 2 Meaningful use criteria. The CTPR is a subset of the USWR data. All patient data from all participating outpatient clinics are transmitted to the USWR where it is available for benchmarking, PQRS and other initiatives. Data used for effectiveness research is HIPAA de-identified. These data are derived from structured language entries directly transmitted from electronic health records which also link to billing and charge documents once practitioners sign and lock charts, confirming the veracity of data entries.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving cellular and tissue based products

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients seen at participating hospital based outpatient wound centers to whom CTPs are applied
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Healing | 12 months
  Healing or wound closure by wound type and stratified by Wound Healing Index

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Wound Care Clinic, The Woodlands, Texas, United States